CLINICAL TRIAL: NCT05062187
Title: Lower Extremity in Hemiparetic Proprioception Sensory and Functionality: A Comparative Study
Brief Title: Lower Extremity Proprioception Sensory and Functionality in Hemiparetic
Status: Completed | Type: Observational
Sponsor: Istanbul Aydın University (Other)
Collaborators: Pamukkale University (Other)
Responsible Party: Principal Investigator, Seref Duhan Altug, PT, Istanbul Aydın University
Other Study IDs: E-60116787-020-78427
Record Dates: First submitted 2021-09-21; First posted 2021-09-30 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Hemiparesis Proprioceptive Disorders Gait, Hemiplegic, Healthy Individual, Comparative Study

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Proprioseption in hemiparetics: Proprioception on balance and gait functions in hemiparetic individuals
  Interventions: Other: Proprioseption in hemiparetics
- Healthy Individual: Proprioception on balance and gait functions in healthy individuals
  Interventions: Other: Proprioseption in hemiparetics

INTERVENTIONS:
Other: Proprioseption in hemiparetics — Proprioception on balance and gait functions in hemiparetic individuals

SUMMARY:
The loss of sensorial feedback causes gait impairment in hemiparesis. The studies show that proprioceptive impairment of knee is related to falling in these patients. The aim of this study is to investigate the effects of proprioception on balance and gait functions in hemiparetic individuals.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 20-65 and discharged from the hospital,
* Diagnosed with hemiparesis at least 4 weeks ago,
* First time and unilateral hemiparesis,
* Modified Rankin Score ≤ 3,
* Hodkinson Mental Test ≥ 6,
* Individuals who agree to receive treatment will be included in the study.

Exclusion Criteria:

* Having vision and hearing problems,
* Having other accompanying neurological, psychiatric and/or orthopedic problems other than hemiparesis,
* Medically unstable,
* Diseases that will affect the lower extremity sense,
* Individuals with open wounds, circulation problems, and skin lesions in the area to be treated will be excluded from the study.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hemiparetic individuals Healthy individuals
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-06-13 (Actual); Study Completion 2022-07-13 (Actual)

PRIMARY OUTCOMES:
Sensorial Assessment-1 | 2 minutes
  Semmes-Weinstein Monoflament
Sensorial Assessment-2 | 2 minutes
  Position test for lower extremity
Sensorial Assessment-3 | 2 minutes
  Kinestesia (Electrogoniometer)
Balance assessment | 30 second
  Static balance via SportKAT-550
Gait parameters | 1 minute
  BTS G-Walk Spatiotemporal gait parameters

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Aydın University, Istanbul, Turkey (Türkiye)